CLINICAL TRIAL: NCT01453153
Title: A Phase 1b/2 Multicenter, International, Randomized, Double Blind, Placebo-Controlled, Study of Gemcitabine Combined With PEGPH20 Compared to Gemcitabine Combined With Placebo in Patients With Stage IV Previously Untreated Pancreatic Cancer
Brief Title: Study of Gemcitabine + PEGPH20 vs Gemcitabine Alone in Stage IV Previously Untreated Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Halo-109-201
Record Dates: First submitted 2011-10-13; First posted 2011-10-17 (Estimated); Results first posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-10

CONDITIONS: Stage IV Pancreatic Cancer
Keywords: pancreatic; Cancer; Stage IV; untreated
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Gemcitabine; PEGPH20; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine (Active Comparator): Gemcitabine + Placebo
  Interventions: Drug: Gemcitabine; Drug: Placebo
- PEGPH20 (Experimental): PEGPH20+Gemcitabine
  Interventions: Drug: Gemcitabine; Drug: PEGPH20

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m2 given IV one time a week (Cycle 1: 7 weeks on treatment, 1 week off treatment; Cycle 2+: 3 Weeks on treatment, 1 week off treatment)
  Other Names: Gemzar
Drug: PEGPH20 — (Cycle 1: 7 weeks on treatment/1 week off treatment; Cycle 2+: 3 Weeks on treatment/1 week off treatment). Doses start at 1.0 mcg/kg and modified until recommended Phase 2 dose is determined. Treatment continues until occurrence of significant treatment-related toxicity, progressive disease, or discontinuation criteria are met
  Other Names: PEGylated Recombinant Human Hyaluronidase
  Arms: PEGPH20
Drug: Placebo — (Cycle 1: 7 weeks on treatment/1 week off treatment; Cycle 2+: 3 Weeks on treatment/1 week off treatment).
  Other Names: Saline
  Arms: Gemcitabine

SUMMARY:
Phase 1B: Open label (all patients receive PEGPH20+gemcitabine), dose escalation, safety and tolerability study to determine the safe dose of PEGPH20 to use in combination with gemcitabine in Stage IV previously untreated pancreatic cancer patients.

Phase 2: Randomized, double blind study to compare the effect of overall survival of gemcitabine plus PEGPH20 vs gemcitabine plus placebo in Stage IV previously untreated pancreatic cancer patients.

DETAILED DESCRIPTION:
PEGPH20 is a PEGylated version of human recombinant PH20 hyaluronidase that, in preclinical studies, has been shown to remove HA from the extracellular matrix surrounding tumor cells by depolymerizing this substrate. 87% of pancreatic ductal adenocarcinomas (PDA) overexpress HA. PDA tumor tissue may be especially sensitive to the HA-degradation properties of PEGPH20 and thus more responsive to the cytotoxic effects of a given dose of gemcitabine. Modifying the extracellular environment to increase the penetration and efficacy of anti-cancer agents represents a novel approach to treating pancreatic cancer and may provide important therapeutic outcomes in patients with Stage IV Previously Untreated Pancreatic Cancer.

This Phase 1B/2 study will assess safety, tolerability, treatment effect, and various PK/PD endpoints.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with histologically confirmed Stage IV adenocarcinoma of the pancrease previously untreated for metastatic disease
* One or more metastatic tumors measurable on CT scan per RECIST 1.1 criteria
* Life expectancy of at least 3 months
* Signed, written IRB/EC-approved informed consent
* A negative serum pregnancy test, if female

Key Exclusion Criteria:

* Known brain metastasis
* New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 12 months
* Active, uncontrolled bacterial, viral, or fungal infection requiring systemic therapy
* Known allergy to hyaluronidase
* Women currently pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy H Zhu, MD, PhD, Study Director — Halozyme Therapeutics
Locations (12):
- United States (8):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - California Pacific Medical Center, San Francisco, California
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - UMDNJ - New Jersey Medical School, Newark, New Jersey
  - NSLIJ Health System, Monter Cancer Center, New Hyde Park, New York
  - Mount Sinai School of Medicine, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Seattle Cancer Care Alliance, Seattle, Washington
- Russia (4):
  - Chelyabinsk Regional Clinical Oncology Center, Chelyabinsk
  - Russian Oncological Research Center n.a. N.N. Blokhin, Moscow
  - Medical Radiological Research Center, Obninsk
  - Omsk Regional Budget Medical Institution, Omsk

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was to consist of a Phase 1b and a randomized Phase 2 study. However, the randomized Phase 2 study was not conducted due to a change to the standard-of-care chemotherapy treatment to be used in combination with PEGylated Recombinant Human Hyaluronidase PH20 (PEGPH20).
Groups:
- PEGPH20 1.0 μg/kg: Participants received PEGylated Recombinant Human Hyaluronidase PH20 (PEGPH20) 1.0 micrograms per kilogram (μg/kg). PEGPH20 was administered twice weekly for 4 consecutive weeks and then once weekly for the next 3 weeks during Cycle 1. For each cycle thereafter, PEGPH20 was administered once weekly for 3 consecutive weeks. Participants received gemcitabine 1000 milligrams per meters squared (mg/m^2) administered via intravenous (IV) infusion. Before the Recommend Phase 2 Dose (RP2D) was established, gemcitabine was administered 2 hours after the second dose of PEGPH20 during Weeks 1 to 4 of Cycle 1 and on the same day as PEGPH20 during each week thereafter. After the RP2D was established, gemcitabine was administered within 24 hours after the first dose of PEGPH20 during Weeks 1 to 4 of Cycle 1 and 2 to 24 hours after each PEGPH20 dose thereafter. Dexamethasone was administered approximately 1 hour prior to and 8 to 12 hours after PEGPH20 dosing.
- PEGPH20 1.6 μg/kg: Participants received PEGPH20 1.6 μg/kg. PEGPH20 was administered twice weekly for 4 consecutive weeks and then once weekly for the next 3 weeks during Cycle 1. For each cycle thereafter, PEGPH20 was administered once weekly for 3 consecutive weeks. Participants received gemcitabine 1000 mg/m^2 administered via IV infusion. Before the RP2D was established, gemcitabine was administered 2 hours after the second dose of PEGPH20 during Weeks 1 to 4 of Cycle 1 and on the same day as PEGPH20 during each week thereafter. After the RP2D was established, gemcitabine was administered within 24 hours after the first dose of PEGPH20 during Weeks 1 to 4 of Cycle 1 and 2 to 24 hours after each PEGPH20 dose thereafter. Dexamethasone was administered approximately 1 hour prior to and 8 to 12 hours after PEGPH20 dosing.
- PEGPH20 3.0 μg/kg: Participants received PEGPH20 3.0 μg/kg. PEGPH20 was administered twice weekly for 4 consecutive weeks and then once weekly for the next 3 weeks during Cycle 1. For each cycle thereafter, PEGPH20 was administered once weekly for 3 consecutive weeks. Participants received gemcitabine 1000 mg/m^2 administered via IV infusion. Before the RP2D was established, gemcitabine was administered 2 hours after the second dose of PEGPH20 during Weeks 1 to 4 of Cycle 1 and on the same day as PEGPH20 during each week thereafter. After the RP2D was established, gemcitabine was administered within 24 hours after the first dose of PEGPH20 during Weeks 1 to 4 of Cycle 1 and 2 to 24 hours after each PEGPH20 dose thereafter. Dexamethasone was administered approximately 1 hour prior to and 8 to 12 hours after PEGPH20 dosing.
Period: Overall Study
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Started | 4 | 4 | 20
Completed | 0 | 0 | 0
Not Completed | 4 | 4 | 20
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Progressive Disease | 3 | 2 | 16
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Adverse Event | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg | Total
Number analyzed (Participants) | 4 | 4 | 20 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (8.06) | 59.0 (8.72) | 60.3 (13.50) | 58.7 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 10 | 14
  Male | 2 | 2 | 10 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 4 | 18 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: The safety and tolerability profile of PEGPH20 used in combination with gemcitabine was assessed by measuring the number of participants with a DLT during the dose-escalation phase of the study. A DLT was defined as any treatment-emergent National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE), Version 4.0, Grade 3 or greater event occurring within the first 4 weeks of treatment that was considered related to PEGPH20. Any PEGPH20 treatment-related AE that resulted in a drug interruption or reduction might have been considered a DLT at the Investigator's or Sponsor's discretion. Hypersensitivity/infusion reactions related to PEGPH20 dosing were not considered DLTs.
Time Frame: first 4 weeks of Cycle 1
Population: The DLT Evaluable Population: all participants enrolled during the dose escalation portion of the study who received at least 6 of 8 planned doses of PEGPH20 and 3 of 4 doses of gemcitabine in the first 4 weeks or had a DLT in the first 4 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 4 | 4 | 6
Participants | 0 | 0 | 0

2. Primary Outcome: Recommended Phase 2 Dose (RP2D)
Description: The safety and tolerability profile of PEGPH20 used in combination with gemcitabine was assessed by determining the RP2D, the highest dose level at which no more than 1 of 6 evaluable participants experienced a DLT in the first 4 weeks of treatment (considered a safe dose). The RP2D was determined based on review of safety and pharmacokinetic (PK) data from participants enrolled during the dose-escalation phase of the study.
Time Frame: first 4 weeks of Cycle 1
Population: as for outcome 1
Measure: Number; unit: micrograms per kilogram (μg/kg)
Groups:
- PEGPH20 Plus Gemcitabine: Participants received PEGPH20 1.0, 1.6, and 3.0 μg/kg. PEGPH20 was administered twice weekly for 4 consecutive weeks and then once weekly for the next 3 weeks during Cycle 1. For each cycle thereafter, PEGPH20 was administered once weekly for 3 consecutive weeks. Participants received gemcitabine 1000 mg/m^2 administered via IV infusion. Gemcitabine was administered 2 hours after the second dose of PEGPH20 during Weeks 1 to 4 of Cycle 1 and on the same day as PEGPH20 during each week thereafter. Participants received dexamethasone 4 or 8 mg orally, via intramuscular injection, or via IV injection. Dexamethasone (4 to 8 mg) was administered approximately 1 hour prior to and 8 to 12 hours after PEGPH20 dosing.
Arm/Group | PEGPH20 Plus Gemcitabine
Number analyzed (Participants) | 14
micrograms per kilogram (μg/kg) | 3.0

3. Secondary Outcome: Observed Maximum Plasma Concentration (Cmax) Following Single PEGPH20 Doses
Description: Cmax is defined as the observed maximum plasma concentration after the first dose. Blood samples were collected for pharmacokinetic assessment.
Time Frame: Cycle 1, Week 1, Day 1: First visit: predose; 15 minutes, 1, 2, 4, and 24 hours post-PEGPH20 dosing; all other visits: pre-PEGPH20 dose, 1 to 2 hours post-PEGPH20 dose, and immediately after the dose of gemcitabine (on the days gemcitabine was given)
Population: Intent-to-Treat Population: all enrolled participants
Measure: Mean (Standard Deviation); unit: units per milliliter
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 4 | 4 | 20
units per milliliter | 0.604 (0.438) | 1.54 (0.491) | 3.18 (1.28)

4. Secondary Outcome: Cmax Following Twice-weekly PEGPH20 Doses for 3 Consecutive Weeks
Description: Cmax is defined as the observed maximum plasma concentration after the first dose. Blood samples were collected for pharmacokinetic assessment. The 24-hour sample collected at the first visit was optional.
Time Frame: Cycle 1, Week 4, Day 1: First visit: predose; 15 minutes, 1, 2, 4, and 24 hours post-PEGPH20 dosing; all other visits: pre-PEGPH20 dose, 1 to 2 hours post-PEGPH20 dose, and immediately after the dose of gemcitabine (on the days gemcitabine was given)
Population: Intent-to-Treat Population: all enrolled participants. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units per milliliter
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 3 | 4 | 12
units per milliliter | 1.08 (0.0878) | 2.40 (0.542) | 3.98 (1.16)

5. Secondary Outcome: Last Measurable Observed Plasma Concentration (Cmin) Following Single PEGPH20 Doses
Description: Blood samples were collected for pharmacokinetic assessment.
Time Frame: as for outcome 3
Population: Intent-to-Treat Population. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units per milliliter
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 3 | 4 | 20
units per milliliter | 0.626 (0.0607) | 0.651 (0.155) | 0.864 (0.375)

6. Secondary Outcome: Cmin Following Twice-weekly PEGPH20 Doses for 3 Consecutive Weeks
Description: Blood samples were collected for pharmacokinetic assessment. The 24-hour sample collected at the first visit was optional.
Time Frame: as for outcome 4
Population: Intent-to-Treat Population. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Units per milliliter
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 3 | 4 | 12
Units per milliliter | 0.572 (0.0781) | 0.976 (0.568) | 1.52 (0.767)

7. Secondary Outcome: Time to Reach Cmax (Tmax) Following Single PEGPH20 Doses
Description: Blood samples were collected for pharmacokinetic assessment.
Time Frame: as for outcome 3
Population: Intent-to-Treat Population. Only those participants with available data were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 3 | 4 | 20
hours | 0.250 [0.180 to 0.330] | 0.250 [0.250 to 1.15] | 0.420 [0.330 to 2.17]

8. Secondary Outcome: Tmax Following Twice-weekly PEGPH20 Doses for 3 Consecutive Weeks
Description: as for outcome 6
Time Frame: as for outcome 4
Population: Intent-to-Treat Population. Only those participants with available data were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 3 | 4 | 12
hours | 0.330 [0.320 to 0.330] | 0.325 [0.250 to 2.08] | 0.420 [0.420 to 2.15]

9. Secondary Outcome: Apparent Half-life (t1/2) Following Single PEGPH20 Doses
Description: The apparent half-life calculated by ln(2)/λ, where λ was the rate constant for the log-linear portion of the terminal phase. A minimum of 3 values in the postdistribution phase of the plasma concentration-time curve were required for calculation of λ. Blood samples were collected for pharmacokinetic assessment. t1/2 is expressed as harmonic mean and pseudo standard deviation.
Time Frame: as for outcome 3
Population: Intent-to-Treat Population. Only those participants with available data were analyzed. t1/2 values were not calculated for the 1.0 μg/kg dose because there were insufficient data points in the profiles due to low concentrations.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 0 | 2 | 18
hours |  | 18.6 (0.255) | 8.24 (8.03)

10. Secondary Outcome: t1/2 Following Twice-weekly PEGPH20 Doses for 3 Consecutive Weeks
Description: The apparent half-life calculated by ln(2)/λ, where λ was the rate constant for the log-linear portion of the terminal phase. A minimum of 3 values in the postdistribution phase of the plasma concentration-time curve were required for calculation of λ. Blood samples were collected for pharmacokinetic assessment. The 24-hour sample collected at the first visit was optional. t1/2 is expressed as harmonic mean and pseudo standard deviation.
Time Frame: as for outcome 4
Population: Intent-to-Treat Population. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 3 | 2 | 9
hours | 5.60 (3.08) | 19.5 (7.75) | 10.7 (4.06)

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Measurable Plasma Concentration (AUC0-T) Following Single PEGPH20 Doses
Description: Blood samples were collected for pharmacokinetic assessment. AUC0-T was calculated by the linear trapezoidal rule.
Time Frame: as for outcome 3
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: Units*hour/milliliter
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 4 | 4 | 20
Units*hour/milliliter | 1.39 (1.57) | 13.6 (11.8) | 31.5 (18.0)

12. Secondary Outcome: AUC0-T Following Twice-weekly PEGPH20 Doses for 3 Consecutive Weeks
Description: Blood samples were collected for pharmacokinetic assessment. The 24-hour sample collected at the first visit was optional. AUC0-T was calculated by the linear trapezoidal rule.
Time Frame: as for outcome 4
Population: Intent-to-Treat Population. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Units*hour/milliliter
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 3 | 4 | 12
Units*hour/milliliter | 2.99 (0.607) | 21.5 (11.9) | 35.2 (23.5)

13. Secondary Outcome: Plasma Hyaluronan (HA) Concentration at Baseline and After PEGPH20 Administration
Description: The pharmacodynamic activity of PEGPH20 was evaluated by measuring plasma concentrations of HA after PEGPH20 dosing. Peak HA concentrations are the highest concentrations measured after a single dose of PEGPH20. HA samples were collected in Cycle 1 at the following time points: 1) Week 1/Day 1 (first visit) and Week 4 (first visit): predose and 15 minutes, 1, 2, 4, and 24 hours post-PEGPH20 dosing (24-hour sample optional for Week 4); 2) all other visits in Cycle 1: pre-PEGPH20 dose, 1 to 2 hours post-PEGPH20 dose, and immediately after the dose of gemcitabine (on the days gemcitabine was given). HA samples were collected in Cycles 2+ at the following time points: Week 3 of each cycle pre-PEGPH20 dose and 1 to 2 hours post-PEGPH20 dose.
Time Frame: Baseline; post-Baseline (average treatment duration of 94.6 days)
Population: Intent-to-Treat Population. This study was to consist of a Phase 1b and a randomized Phase 2 study. However, the randomized Phase 2 study was not conducted due to a change to the standard-of-care chemotherapy treatment to be used in combination with PEGPH20.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 4 | 4 | 20
nanograms per milliliter
  Baseline | 123.7 (137.6) | 982.3 (1370) | 164.7 (139.6)
  After PEGPH20 administration | 7288 (10027) | 27818 (25866) | 128411 (126357)

14. Secondary Outcome: H-scores, as an Assessment of HA Staining Changes in Tumor Biopsies
Description: An H-score approach methodology was developed and used to analyze staining in the tumor pericellular regions and the stroma separately. The H-score calculation was the sum of the products of the percentage of positive staining areas and the staining intensity (0, 1, 2 or 3), and ranged from 0 to 300. For example: [90% * 1 (weak)] + [10% * 2 (moderate)] + [0% * 3 (strong)] = 110. A score of 0 represents the absence of expression, and an H-score of 300 represents maximum expression. A larger decrease in H-score correlated with a greater target engagement of PEGPH20. As HA is a secreted protein, the scoring was performed in the immediate areas surrounding tumor (pericellular areas) as well as in stroma.
Time Frame: Screening; Cycle 1 Week 7
Population: Intent-to-Treat Population. Only 1 participant had a screening and post-treatment specimen that qualified for staining. This study was to consist of a Phase 1b and a randomized Phase 2 study. However, the randomized Phase 2 study was not conducted due to a change to the standard-of-care chemotherapy treatment to be used in combination with PEGPH20.
Measure: Number; unit: score on a scale
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 0 | 0 | 1
score on a scale
  Screening pericellular tumor H-score |  |  | 40
  Screening stromal H-score |  |  | 260
  Post-treatment pericellular tumor H-score |  |  | 15
  Post-treatment stromal tumor H-score |  |  | 150

15. Secondary Outcome: Percent Change in in the Maximum Standardized Uptake Value (SUVmax), as an Assessment of Total Lesion Metabolic Activity
Description: PEGPH20's effect on the metabolic activities of the tumor was assessed as the percent change in SUVmax (a measure of total lesion metabolic activity) using fluorodeoxyglucose-positron emission tomography/computed tomography (18F-FDG-PET/CT). Assessment was done for the entire cohort of participants, not per treatment group.
Time Frame: Baseline; up to 32 weeks for each individual participant (end of Cycle 7)
Population: Intent-to-Treat Population. Only those participants with available data were analyzed. This study was to consist of a Phase 1b and a randomized Phase 2 study. However, the randomized Phase 2 study was not conducted due to a change to the standard-of-care chemotherapy treatment to be used in combination with PEGPH20.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- PEGPH20 1.0, 1.6, or 3.0 μg/kg: Participants received PEGylated Recombinant Human Hyaluronidase PH20 (PEGPH20) 1.0, 1.6, or 3.0 micrograms per kilogram (μg/kg). PEGPH20 was administered twice weekly for 4 consecutive weeks and then once weekly for the next 3 weeks during Cycle 1. For each cycle thereafter, PEGPH20 was administered once weekly for 3 consecutive weeks. Participants received gemcitabine 1000 milligrams per meters squared (mg/m^2) administered via intravenous (IV) infusion. Before the Recommend Phase 2 Dose (RP2D) was established, gemcitabine was administered 2 hours after the second dose of PEGPH20 during Weeks 1 to 4 of Cycle 1 and on the same day as PEGPH20 during each week thereafter. After the RP2D was established, gemcitabine was administered within 24 hours after the first dose of PEGPH20 during Weeks 1 to 4 of Cycle 1 and 2 to 24 hours after each PEGPH20 dose thereafter. Dexamethasone was administered approximately 1 hour prior to and 8 to 12 hours after PEGPH20 dosing.
Arm/Group | PEGPH20 1.0, 1.6, or 3.0 μg/kg
Number analyzed (Participants) | 28
percent change
  Cycle 1: number analyzed (Participants) | 5
  Cycle 1 | -36.7 (19.2)
  Cycle 3: number analyzed (Participants) | 4
  Cycle 3 | -43.2 (12.4)
  Cycle 5: number analyzed (Participants) | 3
  Cycle 5 | -39.3 (20.6)
  Cycle 7: number analyzed (Participants) | 2
  Cycle 7 | -41.2 (61.0)

16. Secondary Outcome: Mean Volume Transfer Constant (Ktrans) for Scans Across Tissue Sites
Description: Dynamic control enhanced-magnetic resonance imaging (DCE-MRI) provides a measure of the exchange of small-molecule contrast agents between the intracellular and extracellular spaces. Using a 2-compartment pharmacokinetic model, an estimate of tissue (tumor) perfusion can be obtained by determining the exchange rate constant (Ktrans) of contrast exchange. Ktrans is defined as the volume transfer constant between extravascular/extracellular space to plasma space and is a measure of blood flow, vascular permeability, or both. Mean Ktrans values across scan sites are reported per participant. DCE-MRI was performed before the first dosing visit (Week 1/Day 1), 24 hours after the first dose of PEGPH20 in Cycle 1, and 24 hours after the last dose of PEGPH20 in Cycle 1 (Week 7). Assessment was done for the entire cohort of participants, not per treatment group.
Time Frame: Baseline; 24 hours hours; end of Cycle 1 (Week 7)
Population: ITT Population. DCE-MRI scans were performed for 6 participants. Only participants with data available were analyzed. This study was to consist of a Phase 1b and a randomized Phase 2 study. However, the randomized Phase 2 study was not conducted due to a change to the standard-of-care chemotherapy treatment to be used in combination with PEGPH20.
Measure: Mean (Standard Deviation); unit: milliliters (mL) per minute per 100 mL
Arm/Group | PEGPH20 1.0, 1.6, or 3.0 μg/kg
Number analyzed (Participants) | 6
milliliters (mL) per minute per 100 mL
  Participant 1, Baseline | 0.124 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 1, 24 hours | 0.383 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 1, End of Cycle 1 | NA (NA) — A scan was not performed at this time point.
  Participant 2, Baseline | 0.430 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 2, 24 hours | 0.468 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 2, End of Cycle 1 | NA (NA) — A scan was not performed at this time point.
  Participant 3, Baseline | 0.402 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 3, 24 hours | 0.331 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 3, End of Cycle 1 | NA (NA) — A scan was not performed at this time point.
  Participant 4, Baseline | 0.564 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 4, 24 hours | 0.672 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 4, End of Cycle 1 | 0.646 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 5, Baseline | 0.135 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 5, 24 hours | 0.197 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 5, End of Cycle 1 | 0.133 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 6, Baseline | 0.249 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 6, 24 hours | 0.376 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 6, End of Cycle 1 | 0.078 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.

17. Secondary Outcome: Mean Extravascular-Extracellular Volume Fraction (Ve) for Scans Across Tissue Sites
Description: DCE-MRI provides a measure of the exchange of small-molecule contrast agents between the intracellular and extracellular spaces. Ve is defined as the extravascular-extracellular volume fraction and is a measure of extracellular, extravascular space. Mean Ve values across scan sites are reported per participant. DCE-MRI was performed before the first dosing visit (Week 1/Day 1), 24 hours after the first dose of PEGPH20 in Cycle 1, and 24 hours after the last dose of PEGPH20 in Cycle 1 (Week 7). Assessment was done for the entire cohort of participants, not per treatment group.
Time Frame: Baseline; 24 hours hours; end of Cycle 1 (Week 7)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | PEGPH20 1.0, 1.6, or 3.0 μg/kg
Number analyzed (Participants) | 6
milliliters
  Participant 1, Baseline | 0.162 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 1, 24 hours | 0.327 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 1, End of Cycle 1 | NA (NA) — A scan was not performed at this time point.
  Participant 2, Baseline | 0.671 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 2, 24 hours | 0.386 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 2, End of Cycle 1 | NA (NA) — A scan was not performed at this time point.
  Participant 3, Baseline | 0.481 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 3, 24 hours | 0.389 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 3, End of Cycle 1 | NA (NA) — A scan was not performed at this time point.
  Participant 4, Baseline | 0.458 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 4, 24 hours | 0.788 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 4, End of Cycle 1 | 0.751 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 5, Baseline | 0.380 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 5, 24 hours | 0.395 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 5, End of Cycle 1 | 0.550 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 6, Baseline | 0.355 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 6, 24 hours | 0.825 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.
  Participant 6, End of Cycle 1 | 0.425 (NA) — A standard deviation was not calculated for the mean values across scan sites for single participants.

18. Secondary Outcome: Number of Participants With the Indicated Best Response, Per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1
Description: Target lesions (TLs), complete response (CR): Disappearance of all TLs. Partial response (PR): >=30% decrease in the sum of diameters of TLs, referencing baseline sums. Progressive disease (PD): >= 20% increase in the sum of diameters of TLs, referencing the smallest sum (including baseline sum). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of >=5 mm. (The appearance of >=1 new lesions is considered progression.) Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient to qualify for PD, referencing the smallest sum diameters. For nontarget lesions (NTLs), CR: Disappearance of all NTLs and normalization of tumor marker level. All lymph nodes must be nonpathological in size (short axis <10 mm). Incomplete response/SD: Persistence of >=1 NTLs and/or maintenance of tumor marker level above normal limits. PD: Unequivocal progression of existing NTLs. (The appearance of >=1 new lesions is considered progression.)
Time Frame: up to approximately 2 years 4 months
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 4 | 4 | 20
Participants
  CR | 0 | 0 | 0
  PR | 0 | 2 | 8
  SD | 1 | 2 | 6
  PD | 3 | 0 | 0
  Unknown | 0 | 0 | 6

19. Secondary Outcome: Objective Response Rate
Description: Objective Response Rate is defined as the number of participants with a complete response plus the number of participants with a partial response, per RECIST, Version 1.1. For TLs, CR: Disappearance of all TLs. PR: >=30% decrease in the sum of diameters of TLs, referencing baseline sums. For NTLs, CR: Disappearance of all NTLs and normalization of tumor marker level. All lymph nodes must be nonpathological in size (short axis <10 mm). Incomplete response/SD: Persistence of >=1 NTLs and/or maintenance of tumor marker level above normal limits.
Time Frame: up to approximately 2 years 4 months
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 4 | 4 | 20
Participants | 0 | 2 | 8
Statistical Analysis 1: Comparison: PEGPH20 1.0 μg/kg; Test type: Superiority; percentage of participants = 0, 95% CI 2-sided [0 to 60]
Statistical Analysis 2: Comparison: PEGPH20 1.6 μg/kg; Test type: Superiority; percentage of participants = 50, 95% CI 2-sided [7 to 93]
Statistical Analysis 3: Comparison: PEGPH20 3.0 μg/kg; Test type: Superiority; percentage of participants = 40, 95% CI 2-sided [19 to 64]

20. Secondary Outcome: Disease Control Rate
Description: Disease Control Rate is defined as the sum of the number of participants with a complete response, the number of participants with a partial response, and the number of participants with stable disease per RECIST, Version 1.1. For TLs, CR: Disappearance of all TLs. PR: >=30% decrease in the sum of diameters of TLs, referencing baseline sums. SD: Neither sufficient shrinkage to qualify for PR nor sufficient to qualify for PD, referencing the smallest sum diameters. For NTLs, CR: Disappearance of all NTLs and normalization of tumor marker level. All lymph nodes must be nonpathological in size (short axis <10 mm). Incomplete response/SD: Persistence of >=1 NTLs and/or maintenance of tumor marker level above normal limits.
Time Frame: up to approximately 2 years 4 months
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 4 | 4 | 20
Participants | 1 | 4 | 14
Statistical Analysis 1: Comparison: PEGPH20 1.0 μg/kg; Test type: Superiority; percentage of participants = 25, 95% CI 2-sided [1 to 81]
Statistical Analysis 2: Comparison: PEGPH20 1.6 μg/kg; Test type: Superiority; percentage of participants = 100, 95% CI 2-sided [40 to 100]
Statistical Analysis 3: Comparison: PEGPH20 3.0 μg/kg; Test type: Superiority; percentage of participants = 70, 95% CI 2-sided [46 to 88]

21. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS duration was defined as the time from the first dose of PEGPH20 until objective tumor progression or death. Per RECIST, Version 1.1, for the evaluation of target lesions, progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters. Note: the appearance of 1 or more new lesions is also considered progression. For the evaluation of nontarget lesions, progressive disease is defined as the unequivocal progression of existing nontarget lesions. Note: The appearance of 1 or more new lesions is also considered progression.
Time Frame: from the first dose of PEGH20 until objective tumor progression or death (up to approximately 2 years 4 months)
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 4 | 4 | 20
days | 47.0 [45.0 to 100.0] | 276.0 [47.0 to 276.0] | 113.0 [50.0 to 166.0]

22. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the time of the first dose of PEGPH20 until death.
Time Frame: from the time of the first dose of PEGPH20 until death (up to approximately 2 years 4 months)
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 4 | 4 | 20
days | 109.5 [48.0 to 424.0] | 199.5 [96.0 to 529.0] | 220.0 [123.0 to 370.0]

23. Secondary Outcome: Change From Baseline in Carbohydrate Antigen 19-9 or Sialylated Lewis(a) Antigen (CA19-9)
Description: CA19-9 is a tumor marker. Blood samples (plasma) were collected for CA19-9 evaluations.
Time Frame: up to the end of Cycle 10 (up to Week 44)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units per milliliter (U/ml)
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 4 | 4 | 20
Units per milliliter (U/ml)
  Cycle 1, Week 4, Visit 1: number analyzed (Participants) | 3 | 3 | 14
  Cycle 1, Week 4, Visit 1 | 12897.5 (22345.65) | -7833.9 (13567.21) | -11800.3 (38780.49)
  Cycle 1, Week 8, Visit 1: number analyzed (Participants) | 1 | 2 | 13
  Cycle 1, Week 8, Visit 1 | 0.0 (NA) — The standard deviation cannot be calculated for a single participant. | -1.9 (2.69) | -15464.1 (41440.85)
  Cycle 2, Week 4, Visit 1: number analyzed (Participants) | 1 | 2 | 10
  Cycle 2, Week 4, Visit 1 | 0.0 (NA) — The standard deviation cannot be calculated for a single participant. | -1.2 (1.63) | -16581.0 (50738.98)
  Cycle 3, Week 4, Visit 1: number analyzed (Participants) | 0 | 1 | 8
  Cycle 3, Week 4, Visit 1 |  | 0.0 (NA) — The standard deviation cannot be calculated for a single participant. | -12628.0 (72538.77)
  Cycle 4, Week 4, Visit 1: number analyzed (Participants) | 0 | 1 | 8
  Cycle 4, Week 4, Visit 1 |  | 0.0 (NA) — The standard deviation cannot be calculated for a single participant. | -24089.1 (54120.73)
  Cycle 5, Week 4, Visit 1: number analyzed (Participants) | 0 | 1 | 6
  Cycle 5, Week 4, Visit 1 |  | 0.0 (NA) — The standard deviation cannot be calculated for a single participant. | -27214.3 (64893.40)
  Cycle 6, Week 4, Visit 1: number analyzed (Participants) | 0 | 1 | 3
  Cycle 6, Week 4, Visit 1 |  | 0.0 (NA) — The standard deviation cannot be calculated for a single participant. | -53200.6 (88132.74)
  Cycle 7, Week 4, Visit 1: number analyzed (Participants) | 0 | 1 | 1
  Cycle 7, Week 4, Visit 1 |  | 0.0 (NA) — The standard deviation cannot be calculated for a single participant. | -154964 (NA) — The standard deviation cannot be calculated for a single participant.
  Cycle 8, Week 4, Visit 1: number analyzed (Participants) | 0 | 1 | 1
  Cycle 8, Week 4, Visit 1 |  | 0.0 (NA) — The standard deviation cannot be calculated for a single participant. | -154946 (NA) — The standard deviation cannot be calculated for a single participant.
  Cycle 9, Week 4, Visit 1: number analyzed (Participants) | 0 | 0 | 1
  Cycle 9, Week 4, Visit 1 |  |  | -154940 (NA) — The standard deviation cannot be calculated for a single participant.
  Cycle 10, Week 4, Visit 1: number analyzed (Participants) | 0 | 0 | 1
  Cycle 10, Week 4, Visit 1 |  |  | -154937 (NA) — The standard deviation cannot be calculated for a single participant.

24. Secondary Outcome: Change From Baseline in CA19-9 in Participants With a Baseline Value >=59 U/ml
Description: CA19-9 is a tumor marker. Blood samples (plasma) were collected for CA19-9 evaluations.
Time Frame: up to the end of Cycle 10 (up to Week 44)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
Number analyzed (Participants) | 3 | 2 | 17
U/ml
  Cycle 1, Week 4, Visit 1: number analyzed (Participants) | 2 | 1 | 11
  Cycle 1, Week 4, Visit 1 | 19346.2 (27370.41) | -23500.0 (NA) — The standard deviation cannot be calculated for a single participant. | -15018.9 (43611.09)
  Cycle 1, Week 8, Visit 1: number analyzed (Participants) | 0 | 0 | 11
  Cycle 1, Week 8, Visit 1 |  |  | -18274.5 (44769.87)
  Cycle 2, Week 4, Visit 1: number analyzed (Participants) | 0 | 0 | 8
  Cycle 2, Week 4, Visit 1 |  |  | -20724.4 (56673.61)
  Cycle 3, Week 4, Visit 1: number analyzed (Participants) | 0 | 0 | 6
  Cycle 3, Week 4, Visit 1 |  |  | -16835.7 (85332.54)
  Cycle 4, Week 4, Visit 1: number analyzed (Participants) | 0 | 0 | 7
  Cycle 4, Week 4, Visit 1 |  |  | -27530.1 (57504.01)
  Cycle 5, Week 4, Visit 1: number analyzed (Participants) | 0 | 0 | 5
  Cycle 5, Week 4, Visit 1 |  |  | -32656.8 (71005.52)
  Cycle 6, Week 4, Visit 1: number analyzed (Participants) | 0 | 0 | 2
  Cycle 6, Week 4, Visit 1 |  |  | -79800.9 (106251.1)
  Cycle 7, Week 4, Visit 1: number analyzed (Participants) | 0 | 0 | 1
  Cycle 7, Week 4, Visit 1 |  |  | -154964 (NA) — The standard deviation cannot be calculated for a single participant.
  Cycle 8, Week 4, Visit 1: number analyzed (Participants) | 0 | 0 | 1
  Cycle 8, Week 4, Visit 1 |  |  | -154946 (NA) — The standard deviation cannot be calculated for a single participant.
  Cycle 9, Week 4, Visit 1: number analyzed (Participants) | 0 | 0 | 1
  Cycle 9, Week 4, Visit 1 |  |  | -154940 (NA) — The standard deviation cannot be calculated for a single participant.
  Cycle 10, Week 4, Visit 1: number analyzed (Participants) | 0 | 0 | 1
  Cycle 10, Week 4, Visit 1 |  |  | -154937 (NA) — The standard deviation cannot be calculated for a single participant.

25. Secondary Outcome: Change From Baseline in CA19-9 in Participants Classified as Responders and Non-responders
Description: CA19-9 is a tumor marker. Blood samples (plasma) were collected for CA19-9 evaluations. Responders are defined as participants who had a complete response or partial response, and non-responders are defined as participants who had stable disease, progressive disease, or an unknown tumor response, per RECIST, Version 1.1.
Time Frame: up to the end of Cycle 10 (up to Week 44)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: U/ml
Groups:
- Responders: Participants received PEGylated Recombinant Human Hyaluronidase PH20 (PEGPH20) 1.0, 1.6, or 3.0 micrograms per kilogram (μg/kg). PEGPH20 was administered twice weekly for 4 consecutive weeks and then once weekly for the next 3 weeks during Cycle 1. For each cycle thereafter, PEGPH20 was administered once weekly for 3 consecutive weeks. Participants received gemcitabine 1000 milligrams per meters squared (mg/m^2) administered via intravenous (IV) infusion. Before the Recommend Phase 2 Dose (RP2D) was established, gemcitabine was administered 2 hours after the second dose of PEGPH20 during Weeks 1 to 4 of Cycle 1 and on the same day as PEGPH20 during each week thereafter. After the RP2D was established, gemcitabine was administered within 24 hours after the first dose of PEGPH20 during Weeks 1 to 4 of Cycle 1 and 2 to 24 hours after each PEGPH20 dose thereafter. Dexamethasone was administered approximately 1 hour prior to and 8 to 12 hours after PEGPH20 dosing.
- Non-responders: Participants received PEGPH20 1.0, 1.6, or 3.0 μg/kg. PEGPH20 was administered twice weekly for 4 consecutive weeks and then once weekly for the next 3 weeks during Cycle 1. For each cycle thereafter, PEGPH20 was administered once weekly for 3 consecutive weeks. Participants received gemcitabine 1000 mg/m^2 administered via IV infusion. Before the RP2D was established, gemcitabine was administered 2 hours after the second dose of PEGPH20 during Weeks 1 to 4 of Cycle 1 and on the same day as PEGPH20 during each week thereafter. After the RP2D was established, gemcitabine was administered within 24 hours after the first dose of PEGPH20 during Weeks 1 to 4 of Cycle 1 and 2 to 24 hours after each PEGPH20 dose thereafter. Dexamethasone was administered approximately 1 hour prior to and 8 to 12 hours after PEGPH20 dosing.
Arm/Group | Responders | Non-responders
Number analyzed (Participants) | 10 | 18
U/ml
  Cycle 1, Week 4, Visit 1: number analyzed (Participants) | 10 | 10
  Cycle 1, Week 4, Visit 1 | -15677.1 (45962.74) | 675.7 (15184.14)
  Cycle 1, Week 8, Visit 1: number analyzed (Participants) | 10 | 6
  Cycle 1, Week 8, Visit 1 | -16367.0 (47164.85) | -6227.9 (12527.76)
  Cycle 2, Week 4, Visit 1: number analyzed (Participants) | 8 | 5
  Cycle 2, Week 4, Visit 1 | -21587.2 (53784.34) | 1377.1 (21979.93)
  Cycle 3, Week 4, Visit 1: number analyzed (Participants) | 6 | 3
  Cycle 3, Week 4, Visit 1 | -28752.7 (61783.48) | 23830.5 (78609.44)
  Cycle 4, Week 4, Visit 1: number analyzed (Participants) | 8 | 1
  Cycle 4, Week 4, Visit 1 | -19976.6 (54603.40) | -32900.0 (NA) — The standard deviation cannot be calculated for a single participant.
  Cycle 5, Week 4, Visit 1: number analyzed (Participants) | 6 | 1
  Cycle 5, Week 4, Visit 1 | -22347.6 (65803.24) | -29200.0 (NA) — The standard deviation cannot be calculated for a single participant.
  Cycle 6, Week 4, Visit 1: number analyzed (Participants) | 4 | 0
  Cycle 6, Week 4, Visit 1 | -39900.5 (76719.16) |
  Cycle 7, Week 4, Visit 1: number analyzed (Participants) | 2 | 0
  Cycle 7, Week 4, Visit 1 | -77482.1 (109576.2) |
  Cycle 8, Week 4, Visit 1: number analyzed (Participants) | 2 | 0
  Cycle 8, Week 4, Visit 1 | -77472.8 (109563.0) |
  Cycle 9, Week 4, Visit 1: number analyzed (Participants) | 1 | 0
  Cycle 9, Week 4, Visit 1 | -154940 (NA) — The standard deviation cannot be calculated for a single participant. |
  Cycle 10, Week 4, Visit 1: number analyzed (Participants) | 1 | 0
  Cycle 10, Week 4, Visit 1 | -154937 (NA) — The standard deviation cannot be calculated for a single participant. |

ADVERSE EVENTS:
Description: This study was to consist of a Phase 1b and a randomized Phase 2 study. However, the randomized Phase 2 study was not conducted due to a change to the standard-of-care chemotherapy treatment to be used in combination with PEGPH20.
Arm/Group | PEGPH20 1.0 μg/kg | PEGPH20 1.6 μg/kg | PEGPH20 3.0 μg/kg
All-Cause Mortality (participants affected / at risk) | 4/4 | 4/4 | 17/20
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/4 | 13/20
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEGPH20 1.0 μg/kg (N=4) | PEGPH20 1.6 μg/kg (N=4) | PEGPH20 3.0 μg/kg (N=20)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEGPH20 1.0 μg/kg (N=4) | PEGPH20 1.6 μg/kg (N=4) | PEGPH20 3.0 μg/kg (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 8
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 9
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 2
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1
Eyelid pain (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 3
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 6
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 1
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 1
Lip pain (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 8
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 1
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Tongue discolouration (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 5
Application site rash (General disorders) | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 6
Catheter site erythema (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 1
Chills (General disorders) | 0 | 1 | 0
Early satiety (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 11
Injection site extravasation (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 3 | 2 | 11
Pyrexia (General disorders) | 2 | 2 | 1
Thirst (General disorders) | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 2
Candidiasis (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2
Respiratory rate increased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 2
Weight increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 8
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 12
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal ganglia infarction (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 3
Dysgeusia (Nervous system disorders) | 3 | 0 | 2
Headache (Nervous system disorders) | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1
Anger (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 1 | 1 | 5
Mental status changes (Psychiatric disorders) | 1 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Penile oedema (Reproductive system and breast disorders) | 0 | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 3
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information obtained as a result of this study or during the conduct of this study will be regarded as confidential. The Investigator agrees to use the information for the purpose of carrying out this study and for no other purpose, unless written permission from the sponsor (Halozyme) is obtained.